CLINICAL TRIAL: NCT02454595
Title: An Open Registry to Measure the Impact of Adding Genomic Testing (Prolaris®) on the Treatment Decision Following Biopsy in Newly Diagnosed Prostate Cancer Patients at Intermountain Hospitals
Brief Title: Registry to Measure the Impact of Adding Genomic Testing
Status: Terminated | Type: Observational
Why Stopped: lack of enrollment
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Collaborators: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: URO-006
Record Dates: First submitted 2015-05-04; First posted 2015-05-27 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded (FFPE) tissue from blocks or slides of prostatic adenocarcinoma biopsies.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Registry — Physician will complete a series of four questionnaires to capture the treatment decisions based upon standard clinical-pathological information and with the addition of the result of genomic testing (Prolaris test).
  Other Names: Prolaris

SUMMARY:
This is a prospective open registry to measure the impact on first-line therapy of genomic testing of biopsy tissue from recently diagnosed treatment-naïve patients with early stage localized prostate cancer. Physicians will complete a series of questionnaires. Biopsy tissue will be tested using the Prolaris® genomic test and a relative cancer aggressiveness score will be shared with the physician and the patient.

DETAILED DESCRIPTION:
This is a prospective open registry to measure the impact on first-line therapy of genomic testing of biopsy tissue from recently diagnosed treatment-naïve patients with early stage localized prostate cancer . Physicians, using standard clinical-pathological parameters (PSA, Gleason score, clinical stage and percent positive cores), will complete a questionnaire that will record their recommendation for first-line therapy from among various treatment options. A sample of the biopsy tissue will then be tested using the Prolaris® genomic test and a relative cancer aggressiveness score will be shared with the physician. After reviewing and considering the results of the genomic testing but prior to the patient consult, the physician will then complete a second treatment decision questionnaire and VAS again. The physician will then discuss the recommended treatment plan with the patient and record the agreed treatment plan on a third questionnaire. After the initial treatment has been initiated, the physician or research staff will record the actual treatment administered in the fourth questionnaire (preferably recorded within 3 months of the patient consultation).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (< or equal to 12 months), untreated patients with histologically proven adenocarcinoma of the prostate that have the following characteristics:
* PSA less than or equal to 10 ng/dl and
* Gleason's 7 (4+3 or 3+4) or Gleason's 6 and
* Age greater than 55 years old and
* Clinical Stage T1 or T2
* Clinically localized (no evidence on clinical or imaging studies of advanced disease).
* No hormonal therapy including luteinizing hormone-releasing hormone (LHRH) agonist or antagonist, anti-androgen, estrogens or exogenous androgens, when applicable.

Exclusion Criteria:

- Known history of hypogonadism

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed ( ≤ 6 months), untreated patients with histologically proven adenocarcinoma of the prostate
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2014-11; Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
The impact of genomic test results towards selecting a first-line therapy option for newly diagnosed, localized, prostate cancer patients. | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wenstrup, MD, Study Director — Myriad Genetic Laboratories, Inc.
Locations (1):
- Intermountain Healthcare, Salt Lake City, Utah, United States